CLINICAL TRIAL: NCT01080781
Title: Ephrin B1 Regulation in Human Right Appendage
Acronym: REBORD
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 09 159 02
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Diseases
Keywords: Cardiomyopathy; Ephrin-B1 expression; cell-cell junctions; heart rate variability; right appendage
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — right appendage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: normal pressures in right auricle (<10 mmHg) /and or pulmonary artery (<35 mmHg)
- Group 2: high pressures in right auricle (> 10 mmHg) /and or pulmonary artery (>35 mmHg)

SUMMARY:
* Background : Ephrin-B1 is part of the large Eph/Ephrin system which is involved in cell-cell comunication. The role of Ephrin-B1 has scarcely been studied in adulthood. Our team has shown that this protein is expressed in normal heart in mice and humans. In mice with deletion of the gene encoding Ephrin-B1, we have shown progressive development of dilated cardiomyopathy characterized by dramatic disorganization of cardiac tissue architecture and decreased heart rate variability.
* Purpose: Ephrin-B1 protein was recently identified in human heart but its putative role remains unknown. In knockout mice, deletion of efn gene is associated with abnormalities in cardiac architecture linked to defects in cell-cell tight junctions. From a functional point of view, mice develop a dilated cardiomyopathy and exhibit decreased heart rate variability in the frequency domain. The purpose of this study is to assess if Ephrin-B1 expression is regulated in human heart and if expression level correlates with heart rate variability.
* Abstract: Thirty patients suffering from cardiac disease needing surgery will be included and separated in two groups according to pressure levels in right auricle /and or pulmonary artery. Ephrin-B1 expression will be assessed in right appendages at both the transcriptional (quantitative PCR) and protein (Western blot) levels. Furthermore, the putative relationship between Ephrin-B1 expression and heart rate variability (24 hours ECG recordings) will be investigated.

DETAILED DESCRIPTION:
* Outcomes
* Primary: Expression level of gene encoding Ephrin B1 (quantitative PCR normalized against GAPDH gene expression) on human right appendage biopsies
* Secondary: a/ Expression level of Ephrin B1 protein on human right appendage using Western blot and b/ Heart rate variability in both time and spectral domains
* Study design: Exploratory, monocentric , prospective and comparative. Two groups of 15 patients each, age and sex matched, with or without elevated pressures in right auricles or pulmonary arteries will be included.
* Eligibility criteria:

  * Inclusion criteria: patients needing cardiac surgery and who had both right catheterism and 24 hours ECG recording before inclusion; stable medications for at least 4 weeks; age > 18 years.
  * Exclusion criteria: Patient with pace-maker or atrial fibrillation
* Number of subjects: 30 patients in two groups of 15 patients each.
* Statistical analysis: Qualitative and quantitative variables will be compared using McNemar test and t test respectively. A p value < 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing cardiac surgery and who had both right cardiac catheterism and 24 hours ECG recording before inclusion
* Stable medications for at least 4 weeks

Exclusion Criteria:

* Patient with pace-maker or atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac diseases, right appendage
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Expression level of gene encoding Ephrin-B1 | 1 year
  Expression level of gene encoding Ephrin-B1 (quantitative PCR normalized against GAPDH gene expression) on human right appendage biopsies

SECONDARY OUTCOMES:
Expression level of Ephrin B1 protein | 1year
  Expression level of Ephrin B1 protein on human right appendage using Western blot and b/ Heart rate variability in both time and spectral domains

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Senard, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France